CLINICAL TRIAL: NCT02703012
Title: Pilot Clinical Study on Patient-Specific Adjustment of Ventilator Settings Using Electrical Impedance Tomography in Patients With Acute Respiratory Distress Syndrome
Brief Title: Clinical Application of Electrical Impedance Tomography for Individual Adjustment of Ventilator Settings
Acronym: CLEAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Norbert Weiler, Prof. N. Weiler, University Hospital Schleswig-Holstein
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UKSH-EIT-01
Record Dates: First submitted 2016-02-05; First posted 2016-03-09 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: ARDS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adjustment of ventilator settings by EIT (Experimental): Individual Adjustment of Ventilator settings using an algorithm based on electrical impedance tomography.
  Interventions: Other: Adjustment of ventilator settings by EIT

INTERVENTIONS:
Other: Adjustment of ventilator settings by EIT — Diagnostic maneuvers (change in tidal volume, recruitment maneuvers) will be performed to detect overdistention, tidal recruitment and recruitability. Tidal volume will be reduced if overdistention is detected by EIT. Positive end-expiratory pressure will be increased if tidal recruitment or recruitability are detected.

SUMMARY:
First clinical application of an algorithm for individual adjustment of ventilator settings using electrical impedance tomography.

DETAILED DESCRIPTION:
In patients suffering from early Acute Respiratory Distress Syndrome (ARDS), an algorithm for individual adjustment of positive end-expiratory pressure and tidal volume will be applied. After optimization of ventilator settings according to the ARDS Network protocol, lung stress and strain, driving pressure, respiratory system compliance (Crs), regional ventilation delay and PaO2 / FiO2 ratio will be recorded. Subsequently, ventilator settings will be adjusted using an algorithm aiming at recruitment and avoiding tidal recruitment and overdistension using electrical impedance tomography (EIT). After 4 hours of EIT-based optimization ventilator settings, lung stress and strain, driving pressure, respiratory system compliance (Crs), regional ventilation delay and PaO2 / FiO2 ratio will be recorded again. The results will be compared to the ARDS Network approach.

ELIGIBILITY:
Inclusion Criteria:

* Acute Respiratory Distress Syndrome (according to Berlin Definition)

Exclusion Criteria:

* Hemodynamic Instability (defined as mean arterial pressure < 65 mmHg OR heart rate < 40 / min OR heart rate > 150 / min OR cardiac index < 2.0 l/min/m^2 DESPITE adequate fluid resuscitation and adequate therapy with inotropes and / or vasopressors)
* Thoracic burns or severe skin injuries
* High frequency oscillatory ventilation
* Pregnancy
* Severe chronic obstructive pulmonary disease (GOLD IV)
* Esophageal varices > grade I
* Esophageal resection
* Invasive ventilation prior to study inclusion for more than 72 hours after onset of ARDS
* Inspiratory oxygen requirement > 80%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01; Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-04 (Actual)

PRIMARY OUTCOMES:
Stress | 4 hours
  Percentage of patients with lung stress (defined as trans-pulmonary pressure during an end-inspiratory hold) below 27 mbar after 4 hours of adjustment of ventilator settings with the algorithm.
Strain | 4 hours
  Percentage of patients with lung strain (defined as end-inspiratory lung volume divided by functional residual capacity) below 2.0 after 4 hours of adjustment of ventilator settings with the algorithm.

SECONDARY OUTCOMES:
Compliance | 4 hours
  Respiratory system compliance (defined as expiratory tidal volume divided by driving pressure) will be measured after 4 hours of adjustment of ventilator settings with the algorithm
Driving Pressure | 4 hours
  Driving Pressure (defined as difference between airway plateau pressure and positive end-expiratory pressure) will be measured after 4 hours of adjustment of ventilator settings with the algorithm
Standard Deviation of regional ventilation delay | 4 hours
  Standard Deviation of regional ventilation delay, (as described in the publication of Muders et al, Crit Care Med Vol. 40, pp 903-911, 2012) will be measured after 4 hours of adjustment of ventilator settings with the algorithm
PaO2 / FiO2 Ratio | 4 hours
  The ratio between arterial partial pressure of oxygen (PaO2) and fraction of inspired oxygen (FiO2) will be measured after 4 hours of adjustment of ventilator settings with the algorithm

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Schleswig Holstein, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Becher T, Buchholz V, Hassel D, Meinel T, Schadler D, Frerichs I, Weiler N. Individualization of PEEP and tidal volume in ARDS patients with electrical impedance tomography: a pilot feasibility study. Ann Intensive Care. 2021 Jun 2;11(1):89. doi: 10.1186/s13613-021-00877-7. PMID 34080074